CLINICAL TRIAL: NCT06776432
Title: A Phase 2A Double-Blind Randomized, Controlled, Dose Escalation, Parallel- Arm, Safety and Efficacy Study of Sivopixant, Acetazolamide and SASS-001 in Sleep Apnea
Brief Title: Safety and Efficacy Study of Sivopixant, Acetazolamide and SASS-001 in Sleep Apnea
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shionogi Apnimed Sleep Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SVA-SAS-201
Record Dates: First submitted 2025-01-03; First posted 2025-01-15 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Sleep Apnea
Keywords: sleep apnea; obstructive sleep apnea; central sleep apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Sleep Apnea, Central | interventions — sivopixant; Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part A: Sivopixant (Active Comparator): Participants will receive sivopixant oral tablets once daily at bedtime for 17 days.
  Interventions: Drug: Sivopixant
- Placebo (Placebo Comparator): Participants will receive placebo to match the study drug during the 17 days of Part A followed by 13 days of Part B.
  Interventions: Drug: Placebo
- Part B I: Acetazolamide (Active Comparator): After completing Part A, participants will receive acetazolamide oral tablets once daily at bedtime for 3 days.
  Interventions: Drug: Acetazolamide
- Part B II: SASS-001 (Active Comparator): After completing Part B I, participants will receive SASS-001 oral tablets once daily at bedtime for 10 days.
  Interventions: Drug: SASS-001

INTERVENTIONS:
Drug: Sivopixant — Administered as specified in the treatment arm
  Arms: Part A: Sivopixant
Drug: Placebo — Administered as specified in the treatment arm.
  Arms: Placebo
Drug: Acetazolamide — Administered as specified in the treatment arm
  Arms: Part B I: Acetazolamide
Drug: SASS-001 — Administered as specified in the treatment arm
  Arms: Part B II: SASS-001

SUMMARY:
The primary purpose of this study is to evaluate the effectiveness of sivopixant, acetazolamide and SASS-001 in adults with sleep apnea with a central component.

ELIGIBILITY:
Inclusion Criteria:

To enroll, subjects need to have a previous diagnosis of at least one or more of the following comorbidities:

* Stable heart failure with reduced ejection fraction (NYHA class 1-3 inclusive) with or without atrial fibrillation
* Heart failure with preserved ejection fraction (NYHA class 1-3 inclusive) and hypertension (BP>120/80 mmHg at screening visit despite the treatment with ≥2 antihypertensives) with or without atrial fibrillation
* Persistent atrial fibrillation (continuous and sustained for more than 7 days, rate controlled with resting HR<100bpm)1 without heart failure
* History of primary (essential) hypertension with BP at screening visit >130/80 mmHg despite the treatment with >2 antihypertensives
* Evidence of complex sleep apnea (CPAP-emergent central sleep apnea with documented CAI>5 events/h on CPAP within 1 year from screening)

Standard care for heart failure and atrial fibrillation for at least 3 weeks before the screening visit

OSA measures Average ODI4 between 7 and 55 events/h, inclusive, and average SpO2 ≥88% from continuous home pulse oximetry recordings at screening.

AHI4 (Hypopneas defined by 4% oxygen desaturation) of >10 to ≤60 events/h

1. At minimum of 25% central or mixed apneas (as proportion of total apneas) with a minimum of 2.5 central or mixed apneas/hour of sleep
2. OR evidence of clear Cheyne-Stokes breathing pattern during the baseline PSG (regardless of central apnea component).
3. OR evidence of OSA with LGn >0.5 at the baseline PSG (regardless of central apnea component) Average SpO2 during sleep ≥88%

Weight BMI between 18.5 and 40 kg/m2 for men, or 42 kg/m2 for women, inclusive

Male participants If male and sexually active with female partner(s) of childbearing potential, participant must agree, from Study Day 1 through 1 week after the last dose of study drug, to practice the protocol specified contraception. Male participants must refrain from donating sperm for the duration of the study and for 3 months after the last dose of study treatment.

Female participants If a woman of childbearing potential (WOCBP), the participant must agree, from Study Day 1 through 1 week after the last dose of study drug, to practice the protocol specified contraception. All WOCBP must have negative result of a serum pregnancy test performed at screening.

If female and of non-childbearing potential, the participant must be either postmenopausal or permanently sterile (e.g. bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

Informed Consent Participant voluntarily agrees to participate in this study and signs an Institutional Review Board (IRB)-approved informed consent prior to performing any of the Screening Visit procedures.

Participant must be able to understand the nature of the study and must have the opportunity to have any questions answered.

Patients currently using PAP will be eligible for inclusion in the study if they express willingness to discontinue treatment for a minimum of 7 days before baseline SpO2 assessments, until the study completion.

Exclusion criteria Vital signs and symptoms

Sustained SpO2<93% during wakefulness or mean SpO2<88% during sleep, calculated from PSG at screening

Dyspnea at rest or patients with heart failure class IV NYHA

Blood pressure <90/50 mmHg or >160/100 mmHg at V1.

Medical Conditions Recent (<3 months) episode of acute myocardial infarction or acute decompensated heart failure.

History of stroke.

History of sustained ventricular tachyarrhythmias or other severe arrhythmias without defibrillator implanted.

Heart failure primarily caused by valvular, post-partum cardiomyopathy or active myocarditis

History of obesity-hypoventilation syndrome or respiratory disturbance due to opioids.

History of bronchiectasis and uncontrolled asthma.

History of severe chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) <50% of predicted (European Respiratory Society criteria)

Started treatment with β-blockers <3 months before screening. Patients not taking β-blockers or taking β-blockers for >3 months can be enrolled.

Narcolepsy, restless leg syndrome requiring medication, REM sleep behavior disorder.

Pronounced anatomical abnormalities of upper airway (adenoid vegetations, grade ≥3 tonsillar hypertrophy, etc.), pronounced micrognathia, or pronounced incomplete development of the lower jaw.

History of schizophrenia, schizoaffective disorder or bipolar disorder according to Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) or International Classification of Disease tenth edition criteria.

Medically unexplained positive screen for drugs of abuse (excluding THC/marijuana) or history of substance use disorder as defined in DSM-V within 24 months prior to Screening Visit.

A significant illness or infection requiring medical treatment in the past 30 days as determined by investigator.

Clinically significant cognitive dysfunction as determined by investigator.

Women who are pregnant or nursing.

History of kidney stones

Prior/Concomitant Therapy Participants with a history of using devices for OSA treatment, including CPAP, oral or nasal devices, or positional devices, may enroll as long as the devices have not been used for at least 1 week before the baseline SpO2 assessments and are not used during participation in the study (through V7). Patients that are non-compliant to CPAP (less than 4hr/night for 5 days/week) can be enrolled, as well as patients who are naïve to PAP and patients who discontinued PAP previously. PAP compliant patients cannot be enrolled.

History of chronic oxygen therapy.

Concomitant use of medications from the list of disallowed medications.

Prior/Concurrent Clinical Study Experience Use of another investigational agent within 30 days or 5 half-lives, whichever is longer, prior to dosing.

Diagnostic Assessments Hepatic cirrhosis, hepatictransaminases > 2X the upper limit of normal (ULN), total bilirubin >1.5X ULN (unless confirmed Gilbert syndrome), estimated glomerular filtration rate < 40 ml/min.

Participants with reduced sodium and/or potassium blood serum levels.

Participants with suprarenal gland failure.

Participants with hyperchloremic acidosis.

Other Exclusions:

Night- or shift-work sleep schedule which causes the major sleep period to be during the day.

Employment as a commercial driver or operator of heavy or hazardous equipment.

Typically smoking more than 10 cigarettes or 2 cigars per day, or inability to abstain from smoking during overnight PSG visits.

Unwilling to use specified contraception.

History of regular alcohol consumption of more than 14 standard units per week (males) or more than 7 standard units per week (females), or unwillingness to limit alcohol consumption to no greater than 2 units/day (males), 1 unit per day (females). Alcohol is not to be consumed within 3 hours of bedtime or on PSG nights.

Unwilling to agree to limit during the study period caffeinated beverage intake (e.g., coffee, cola, tea) to 400 mg/day or less of caffeine, not to be used within 3 hours of bedtime.

Any condition that in the investigator's opinion would present an unreasonable risk to the participant, including recent (<1 year) motor vehicle accident due to drowsy driving, or which would interfere with their participation in the study or confound study interpretation.

Participant considered by the investigator, for any reason, an unsuitable candidate to receive sivopixant or acetazolamide or unable or unlikely to understand or comply with the dosing schedule or study evaluations.

Allergy to study drugs

• Note: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint - Change in apnea-hypopnea index (SASS-001 arm vs baseline at Visit 7 polysomnography). Scale is minimum -60 to max 60. Lower scores mean improvement from baseline. | up to 6 weeks

SECONDARY OUTCOMES:
Secondary Endpoint - Change in apnea-hypopnea index (Sivopixant alone vs baseline at Visit 5 polysomnography). Scale is minimum -60 to max 60. Lower scores mean improvement from baseline. | up to 6 weeks

OTHER OUTCOMES:
Additional Secondary Endpoint: Change in apnea-hypopnea index (SASS-001 vs Acetazolamide alone - visit 7 vs visit 6 polysomnography). Scale is minimum -60 to max 60. Lower scores mean improvement from baseline. | Two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chief Scientific Officer, Study Director — Shionogi Apnimed Sleep Science
Locations (9):
- United States (9):
  - Altman Clinical and Translational Research Institute (ACTRI), La Jolla, California
  - Teradan Clinical Trials, Brandon, Florida
  - PharmaDev Clinical Research Institute, LLC, Miami, Florida
  - Infinity Medical Research, North Dartmouth, Massachusetts
  - John D. Dingell VA Medical Center, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Intrepid Research, LLC, Cincinnati, Ohio
  - OnSite Clinical Solutions, Rock Hill, South Carolina
  - Huntsville Research Institute LLC, Huntsville, Texas